CLINICAL TRIAL: NCT03293732
Title: A Randomized, Double-blind Phase I Trial to Evaluate the Safety, Tolerability, and Immunogenicity of DCB07010 Adjuvant Given Intranasally at Ascending Dose Levels and Co-administered With Trivalent Inactivated Influenza Virus Antigen
Brief Title: Study of the Safety, Tolerability and Immunogenicity of an Intranasal Influenza Vaccine Administered to Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Advagene Biopharma Co. Ltd. (Industry)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DCB07030-CT-01
Record Dates: First submitted 2017-09-19; First posted 2017-09-26 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Flu, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- HA antigen only (Active Comparator): All subjects in this group received 2 doses of 22.2 μg HA antigens
  Interventions: Biological: HA antigens
- 7.5 μg of DCB07010 (Experimental): All subjects in this group received 7.5 μg of DCB07010 in 22.2 μg HA antigens twice.
  Interventions: Biological: DCB07010; Biological: HA antigens
- 15 μg of DCB07010 (Experimental): All subjects in this group received 15 μg of DCB07010 in 22.2 μg HA antigens twice.
  Interventions: Biological: DCB07010; Biological: HA antigens
- 30 μg of DCB07010 (Experimental): All subjects in this group received 30 μg of DCB07010 in 22.2 μg HA antigens twice.
  Interventions: Biological: DCB07010; Biological: HA antigens
- 45 μg of DCB07010 (Experimental): All subjects in this group received 45 μg of DCB07010 in 22.2 μg HA antigens twice.
  Interventions: Biological: DCB07010; Biological: HA antigens

INTERVENTIONS:
Biological: DCB07010 — A protein based adjuvant originated from prokaryotic organism.
  Arms: 15 μg of DCB07010; 30 μg of DCB07010; 45 μg of DCB07010; 7.5 μg of DCB07010
Biological: HA antigens — HA antigens from three strains of influenza virus ( 7.5 μg of HA each strain).

SUMMARY:
The objectives of this study were to assess the safety and tolerability of DCB07010 when given intranasally at escalating dose levels of 7.5μg, 15μg, 30μg and 45μg, in combination with 22.5μg of influenza HA antigen (7.5μg HA of each of three strains) and to generate sufficient immunogenicity data to enable dose selection for larger and more definitive Phase 2 studies.

This was a single center, double-blind, randomized (2:1), dose-escalation study to assess the safety, tolerability and immunogenicity of 4 different vaccine-adjuvant doses in comparison to influenza HA alone. The 4 treatment cohorts were given DCB07010 in a dose- escalating manner.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking adult aged between 20-40 years old;
2. Physically and mentally healthy subjects as confirmed by an interview, medical history, clinical examination, chest X-rays, ophthalmoscopy, cardiac echo, and electrocardiogram;
3. Body Mass Index (BMI) between 18.5 and 25, inclusive, (BMI will be calculated as weight in kilogram [kg]/height in meters2 [m2]);
4. Normal hematology, biochemistry and urinalysis determinations;
5. Subject is willing and able to comply with study procedures and sign informed consent

Exclusion Criteria:

1. Subject with serious underlying chronic illness;
2. Documented evidence of allergic rhinitis;
3. Subject with acute sinusitis or chronic sinusitis accompanying acute symptoms within 3 days prior to enrollment;
4. Immunosuppressed subjects as result of illness or treatment;
5. Female subject of childbearing potential who:

   * is lactating; or
   * has positive urine pregnancy test at Visit 2 or Visit 3; or
   * refuse to adopt reliable method of contraception during the study;
6. Subject received blood products or immunoglobulin within 3 months prior enrollment;
7. Subjects with long-term use of steroids, including parenteral steroids or high dose inhaled steroids within 28 days prior to enrollment;
8. Subject has received any intranasal medication or nasal topical treatment within 7 days prior to enrollment;
9. Subject has received any investigational agent within 28 days or 5 half- lives, whichever is longer, prior to the first dose of investigational product;
10. Subject has previously experienced anaphylaxis;
11. Subject has allergy to eggs or prior influenza vaccine;
12. Subject with laboratory-confirmed influenza or has been vaccinated against influenza within 6 months prior to enrollment;
13. Subject with acute respiratory illness or administered antibiotics or antivirals within 7 days prior to enrollment;
14. Subject with body temperature high than 38°C within 3 days prior to enrollment;
15. Subject with documented history of Bell's palsy or neurological disorder.
16. Subject with documented history of diarrhea within one month prior to study enrollment
17. A positive test for HIV antibody.
18. Subject has received Chinese medication or herbal medication within 28 days prior to enrollment

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-11-28 (Actual); Primary Completion 2013-03-30 (Actual); Study Completion 2013-09-30 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Titers (GMT) against all three strains of viral antigen | Day=0, 28
  Geometric Mean Titers (GMT) against all three strains of viral antigen after 2 doses of DCB07010 adjuvanted egg-derived vaccines or egg-derived vaccine. The geometric mean titers against all three-vaccine strains were assessed by egg-derived antigen haemagglutination inhibition (HI) assay.
  Statistic tests were two-sided and were set for alpha = 0.05. The purpose of this study was exploratory in safety and the formal statistical analysis was not necessary.

SECONDARY OUTCOMES:
Geometric Mean Ratio (GMR) after 2 dose of vaccines | Day=0, 28
  Geometric Mean Ratio (GMR) after 2 dose of egg-based vaccine and DCB07010-adjuvanted vaccines. Statistic tests were two-sided and were set for alpha = 0.05. The purpose of this study was exploratory in safety and the formal statistical analysis was not necessary.
Seroconversion Rates (SCR) measurements | Day=0, 28
  Seroconversion Rates (SCR) is defined the percentage of subjects with pre-vaccination HI titers < 1:10 and a post-vaccination titer ≥ 1:40 or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer to each of the three vaccine components on Day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Shaun-Chwen Chang, Ph.D., Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan Univserity Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pan SC, Hsieh SM, Lin CF, Hsu YS, Chang M, Chang SC. A randomized, double-blind, controlled clinical trial to evaluate the safety and immunogenicity of an intranasally administered trivalent inactivated influenza vaccine with adjuvant LTh(alphaK): A phase I study. Vaccine. 2019 Mar 28;37(14):1994-2003. doi: 10.1016/j.vaccine.2019.02.006. Epub 2019 Mar 2. PMID 30837170